CLINICAL TRIAL: NCT05192421
Title: A Remotely Delivered, Web-Based Exercise Intervention for Sedentary Adults: Randomized Controlled Pilot Trial
Brief Title: An mHealth Exercise Intervention for Sedentary Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Responsible Party: Principal Investigator, Jackie Kiwata Dawson, PhD, Principal Investigator, California State University, Long Beach
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-240
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Exercise Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level 1 (Active Comparator): Wellness Education
  Interventions: Behavioral: Wellness Education
- Level 2 (Experimental): Wellness Education + Pre-recorded Exercise Videos
  Interventions: Behavioral: Wellness Education; Behavioral: Exercise Videos
- Level 3 (Experimental): Wellness Education + Livestream Exercise Classes
  Interventions: Behavioral: Wellness Education; Behavioral: Livestream Classes

INTERVENTIONS:
Behavioral: Wellness Education — Receive wellness education through a weekly email and web portal content.
Behavioral: Exercise Videos — Receive pre-recorded exercise videos through a weekly email and web portal content.
  Arms: Level 2
Behavioral: Livestream Classes — Receive 3 videoconference group exercise classes per week for 8 weeks.
  Arms: Level 3

SUMMARY:
This pilot trial examines the feasibility and acceptability of a web-based, social networking exercise intervention in improving physical activity behavior in adults who do not perform regular exercise.

DETAILED DESCRIPTION:
Primary Objective To determine the feasibility and acceptability of an 8-week remotely-delivered exercise intervention by conducting a randomized controlled study comparing 3 levels of behavioral engagement.

Secondary Objectives

To compare the effectiveness of 3 levels of web-based interaction on physical activity behavior, physiological training dose, motivation and quality of life. Participants are randomly assigned to 1 of 3 groups:

Level 1 (attention control): Participants receive health educational materials through email and the web portal.

Level 2 (videos): Participants receive health education materials + access to 24 pre-recorded exercise videos.

Level 3 (livestream classes): Participant receive health education materials + livestream exercise classes 3 days/week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Not exceeding 60 total minutes of physical activity per week
* Access to computer or mobile device with high speed internet connection

Exclusion Criteria:

* History of myocardial infarction, angioplasty, coronary artery bypass, cerebrovascular ischemia/stroke, symptomatic congestive heart failure, atrial flutter, unstable angina, or unstable pulmonary disease; pacemaker; history of alcoholism, drug abuse or other psychiatric problems; current use of tricyclic antidepressant or clozapine medications; type 1 diabetes; orthopedic or rheumatologic problems that could impair the ability to walk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Accrual | Up to 1 year
  Measured as the percentage of the eligible target sample enrolled within a 1-year recruitment period.
Retention | Up to 1 month
  Measured as the percentage of participants completing post-intervention assessments
Adherence | Up to 2 months
  Measured as the number sessions completed using activity tracker

SECONDARY OUTCOMES:
Moderate to Vigorous Physical Activity | Up to 2 months
  Amount of time per week spent performing activity >63% maximum heart rate
Resting Heart Rate | Baseline, 2 months
  Average heart rate over a 10 minute period taken while sitting at rest
International Physical Activity Questionnaire (IPAQ) | Baseline, 2 months
  IPAQ estimates weekly moderate to vigorous intensity physical activity
Short Form-36 (SF-36) | Baseline, 2 months
  A 36-item survey that assesses general quality of life status
Profile of Mood States (POMS) | Baseline, 2 months
  A 65-item survey that assesses the participant's mood
Physical Activity Group Questionnaire | Baseline, 2 months
  A 21-item survey that assesses individual and group perceptions of task and social cohesion

CONTACTS AND LOCATIONS:
Locations (1):
- California State University, Long Beach, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson JK, Ede A, Phan M, Sequeira A, Teng HL, Donlin A. Feasibility and Acceptability of a Mobile Health Exercise Intervention for Inactive Adults: 3-Arm Randomized Controlled Pilot Trial. JMIR Form Res. 2024 Aug 9;8:e52428. doi: 10.2196/52428. PMID 39120078